CLINICAL TRIAL: NCT05185830
Title: The Effect Of Interactive Robot on Children's Anxiety, Mobilization and Parental Satisfaction After The Surgery
Brief Title: The Effect Of Interactive Robot on Children's After The Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Collaborators: Koç University (Other)
Responsible Party: Principal Investigator, Sacide Yildizeli Topcu, Assistant Professor, Trakya University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020.17
Record Dates: First submitted 2021-12-21; First posted 2022-01-11 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Pediatric Surgery
Keywords: interactive robot; child; surgery; mobilization; anxiety; parental satisfaction
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Non-Randomized study with control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interactive robot (Experimental): Children in the interactive robot will be mobilized for the first time with interactive robots.
  Interventions: Other: Interactive robots
- Control group (No Intervention): Children in the control group will be mobilized with nurses

INTERVENTIONS:
Other: Interactive robots — Children will mobilize with the interactive robot when control group will mobilize with nurse.
  Arms: Interactive robot

SUMMARY:
This project will be conducted with 5-10-year-old children who will undergo an outpatient surgery in Trakya University Health Research and Application Center at Pediatric Surgery Clinic and their parents. It is reported in the literature that technology-based applications and robot use are promising innovations in reducing pain, anxiety, and fear in children. This was the main starting point in the planning of the study. In this study, by using interactive robot, it was aimed to reduce postoperative mobilization anxiety, to increase frequency / duration of the mobilization and to increase parental satisfaction of the children undergoing outpatient surgery.

DETAILED DESCRIPTION:
The use of interactive robots is expected to reduce the child's anxiety by ensuring that the child is physically, psychologically, and socially optimal. It is foreseen that the child with reduced anxiety will be willing to mobilize with the interactive robot and it will increase the mobilization time and the frequency of the mobilization during the day. Decreasing the anxiety of children and increasing the desire for mobilization will increase the satisfaction of the families.

The study will be conducted with 84 children (42 Experiment + 42 Control) aged 5-10 years. The study was planned as a randomized controlled study. Data will be collected by "Questionnaire Form" and "Child Anxiety Scale-State Anxiety" and Parental Satisfaction Scoring-Visual Analog Scale" and "Mobilization Chart". Families will be informed about the research and before the surgery, families, and children in both groups will be informed about the benefits of mobilization. Two hours after the operation, just before the mobilization, the children in the experimental group will be introduced to the robot, and the children in the control group will be asked to mobilize with their parents.

When the child is first mobilized at the time recommended by the physician for all groups after the surgery, the child's anxiety for mobilization will be assessed using the Child Anxiety Scale (State Anxiety). The mobilization time of the children will be measured by stopwatch and recorded in the Mobilization Schedule together with the frequency of mobilization. Parental Satisfaction Scale- Visual Analogue Scale will be applied to evaluate the satisfaction of the parents towards the application.

ELIGIBILITY:
Inclusion Criteria:

* Undergo day surgery,
* Speaking Turkish,
* Being a volunteer to participate in the study,
* Being 5-10 aged,
* Do not have a visual, auditory, or mental problem and their parents will be included in the research.

Exclusion Criteria:

* No undergo day surgery,
* No Speaking Turkish,
* Not being a volunteer to participate in the study,
* Not being 5-10 aged,
* Have a visual, auditory, or mental problem and their parents will be included in the research.

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2021-01-29 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Anxiety assessment by the Child Anxiety Scale-State Anxiety | Baseline (Before the mobilization)
  The Children's Anxiety Meter assesses children's anxiety and uses before medical procedures. This scale is drawn like a thermometer with a bulb at the bottom and also includes horizontal lines at intervals going up to the top (0-10). This scale ranges from 0 to 10. Higher values represent higher anxiety.
Parental Satisfaction assessment by Parental Satisfaction Scoring-Visual Analog Scale | After the postop children's mobilization up to 6 hours
  Parental Satisfaction Score-Visual Analog Scale is scored as "0-not satisfied at all", "10-very satisfied". It will be used to evaluate the satisfaction of the parents of the children in the whole group towards post-operative nursing care.
Mobilization duration assessment by the Mobilization Chart | walking time at the child's first mobilization up to 6 hours
  The mobilization schedule created by the researchers ensures that the time the child was mobilized on the first and second days after the surgery and the standing/walking time during each mobilization were recorded. The chart will be filled by the nurses. A stopwatch will be used to calculate the standing time. The stand-up period will start with the child getting up from the bed and will end when he/she goes back to bed.
Mobilization frequency assessment by the Mobilization Chart | through study completion, an average of 6 hours
  The mobilization schedule created by the researchers ensures that the time the child was mobilized on the first and second days after the surgery and the standing/walking time during each mobilization were recorded. The chart will be filled by the nurses. A stopwatch will be used to calculate the standing time. The stand-up period will start with the child getting up from the bed and will end when he/she goes back to bed.

CONTACTS AND LOCATIONS:
Overall Officials: Sacide YILDIZELİ TOPÇU, PhD, Principal Investigator — Trakya University
Locations (1):
- Remziye Semerci, Edirne, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol